CLINICAL TRIAL: NCT01984749
Title: A Multicenter, Randomized, Comparative Trial on the Effect of Febuxostat in Preventing Cerebral and Cardiorenovascular Events in Patients With Hyperuricemia
Brief Title: Febuxostat for Cerebral and caRdiorenovascular Events prEvEntion stuDy
Acronym: FREED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Freed Study Group (Other)
Collaborators: Teijin Pharma Limited (Industry)
Responsible Party: Principal Investigator, Hisao Ogawa, Deputy Director General of the hospital, National Cerebral and Cardiovascular Center Hospital, Freed Study Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0078; UMIN000012134 (Registry Identifier: UMIN)
Record Dates: First submitted 2013-10-30; First posted 2013-11-15 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — Febuxostat

ARMS (2):
- Febuxostat treatment group (Experimental): Once daily after breakfast (generally within 30 minutes after eating)
  Interventions: Drug: Febuxostat
- Non-febuxostat treatment group (No Intervention): No febuxostat treatment

INTERVENTIONS:
Drug: Febuxostat — Febuxostat will be taken once daily after breakfast (generally within 30 minutes after eating) but can be taken around the time of breakfast even if no food has been eaten. When the dose is to be increased, the principal or sub-investigator will carry out any required examinations and tests as needed.
  1. The starting dose of the investigational product (febuxostat) will be 10 mg/day.
  2. The dose will be increased to 20 mg/day at Week 4.
  3. The aim is to increase the dose to 40 mg/day at Week 8.
  Arms: Febuxostat treatment group

SUMMARY:
The purpose of this study is to demonstrate the effect of febuxostat in preventing cerebral and cardiorenovascular events in elderly patients with hyperuricemia who are at risk for cerebral and cardiorenovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* (1) Patients 65 years of age or older at enrollment who are able to visit
* (2) Patients with hyperuricemia, who have a serum uric acid level >7.0 mg/dL and <= 9.0 mg/dL (7.0 mg/dL < serum uric acid level <= 9.0 mg/dL) within 2 months prior to enrollment
* (3) Patients at risk for any of the cerebral or cardiorenovascular diseases in i) through iv) below (i) Previous or current history of hypertension (ii) Previous or current history of type 2 diabetes mellitus (iii) Renal disorders (30 mL/min/1.73 m2 <= eGFR < 60 mL/min/1.73 m2 within 3 months prior to enrollment) (iv) Previous history of cerebral or cardiorenovascular disease for more than 3 months prior to enrollment (stroke [cerebral hemorrhage, cerebral infarction, or subarachnoid hemorrhage], coronary artery disease, vascular disease, or cardiac failure)
* (4) Patients who personally give written informed consent to participate in this study

Exclusion Criteria:

* (1) Patients with gouty tophus, or patients with subjective symptoms of gouty arthritis within 1 year prior to enrollment
* (2) Patients with a previous history of hypersensitivity to febuxostat or allopurinol
* (3) Patients with malignant tumors
* (4) Patients with serious kidney disease, Acute kidney disease, nephrotic syndrome, dialysis patients, kidney transplant patients, eGFR < 30 mL/min/1.73 m2 , etc.
* (5) Patients with a previous history of acute coronary syndrome or stroke within 3 months prior to enrollment (cerebral hemorrhage, cerebral infarction, or subarachnoid hemorrhage)
* (6) Patients with a >= 50% increase in serum creatinine within 3 months prior to enrollment
* (7) Patients with severe hypertension characterized by systolic blood pressure >= 180 mmHg or diastolic blood pressure >= 110 mmHg within 3 months prior to enrollment
* (8) Patients with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) 2 or more times the upper limit of normal within 3 months prior to enrollment
* (9) Patients on any of the following medications at enrollment Mercaptopurine hydrate, azathioprine, vidarabine, or didanosine
* (10) Patients who receive any of the following medications for the treatment of hyperuricemia within 1 month prior to enrollment Allopurinol, benzbromarone, probenecid, bucolome, topiroxostat, or febuxostat
* (11) Patients who start, modify the dose of, or discontinue any of the following medications within 1 month prior to enrollment Losartan, irbesartan, fenofibrate, thiazide diuretics, or loop diuretics
* (12) Patients on hormone replacement therapy with estrogen (estrogenic hormone products)
* (13) Patients who have participated in other clinical research (including trials) within 6 months prior to enrollment (non-interventional observational research not excluded)
* (14) Patients otherwise judged by the principal or sub-investigator to be unsuitable for the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-11; Primary Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Development of cerebral or cardiorenovascular events and all deaths | Enrollment through Month 36
  Definition of "cerebral and cardiorenovascular events":
  1. Death due to cerebral or cardiorenovascular disease
  2. New or recurrent cerebrovascular disease (stroke [cerebral hemorrhage, cerebral infarction, subarachnoid hemorrhage, stroke of unknown type], transient ischemic attack
  3. New or recurrent non-fatal coronary artery disease (myocardial infarction and unstable angina pectoris)
  4. Cardiac failure requiring hospitalization
  5. Arteriosclerotic disease requiring hospitalization (aortic aneurysm, aortic dissection, and arteriosclerosis obliterans)
  6. Renal impairment (development of microalbuminuria, progression to overt proteinuria, or overt proteinuria [≥ 300 mg/gCr], confirmed by two consecutive laboratory tests performed after the initiation of study treatments; doubling of serum creatinine level; and progression to ESRD)
  7. New atrial fibrillation (including paroxysmal atrial fibrillation)
  8. Deaths that are not caused by cerebral or cardiorenovascular disease

SECONDARY OUTCOMES:
Occurrence of cerebral or cardiorenovascular event by event | Enrollment through Month 36
Occurrence of cerebral or cardiorenovascular event by serum uric acid level | Enrollment through Month 36
Occurrence of cerebral or cardiorenovascular event by prior history of cerebral or cardiorenovascular disease | Enrollment through Month 36
Serum uric acid level | At screening, at enrollment, at 4, 8, and 12 weeks and 6, 12, 18, 24, 30, and 36 months (or at withdrawal from the study)
Change in serum uric acid level | Enrollment through Week 4
Amount of change and percent change in serum uric acid level | Enrollment through Week 8
Amount of change and percent change in serum uric acid level | Enrollment through Week 12
Amount of change and percent change in serum uric acid level | Enrollment through Month 6
Amount of change and percent change in serum uric acid level | Enrollment through Month 12
Amount of change and percent change in serum uric acid level | Enrollment through Month 18
Amount of change and percent change in serum uric acid level | Enrollment through Month 24
Amount of change and percent change in serum uric acid level | Enrollment through Month 30
Amount of change and percent change in serum uric acid level | Enrollment through Month 36 (or withdrawal from the study)
Percent Achieving serum uric acid level of 6.0mg/dL | Enrollment to completion of study or withdrawal
Estimated glomerular filtration rate (eGFR) | Enrollment, 4, 8, and 12 weeks and 6, 12, 18, 24, 30, and 36 months (or withdrawal from the study)
Amount of change and percent change in eGFR | Enrollment through Week 4
Amount of change and percent change in eGFR | Enrollment through Week 8
Amount of change and percent change in eGFR | Enrollment through Week 12
Amount of change and percent change in eGFR | Enrollment through Month 6
Amount of change and percent change in eGFR | Enrollment through Month 12
Amount of change and percent change in eGFR | Enrollment through Month 18
Amount of change and percent change in eGFR | Enrollment through Month 24
Amount of change and percent change in eGFR | Enrollment through Month 30
Amount of change and percent change in eGFR | Enrollment through Month 36 (or withdrawal from the study)
Urine microalbumin-creatinine ratio | Enrollment, 6, 12, 24, and 36 months (or withdrawal from the study)
Amount of change and percent change in urine microalbumin-creatinine ratio | Enrollment through Month 6
Amount of change and percent change in urine microalbumin-creatinine ratio | Enrollment through Month 12
Amount of change and percent change in urine microalbumin-creatinine ratio | Enrollment through Month 24
Amount of change and percent change in urine microalbumin-creatinine ratio | Enrollment through Month 36 (or withdrawal from the study)
Quantification of urinary protein | Enrollment, 6, 12, 24, and 36 months (or withdrawal from the study)
Amount of change and percent change in quantified urinary protein | Enrollment through Month 6
Amount of change and percent change in quantified urinary protein | Enrollment through Month 12
Amount of change and percent change in quantified urinary protein | Enrollment through Month 24
Amount of change and percent change in quantitative urinary protein | Enrollment through Month 36 (or withdrawal from the study)
Blood pressure (systolic/diastolic) | Enrollment, 6, 12, 18, 24, 30, and 36 months (or withdrawal from the study)
Amount of change and percent change in blood pressure (systolic/diastolic) | Enrollment through Month 6
Amount of change and percent change in blood pressure (systolic/diastolic) | Enrollment through Month 12
Amount of change and percent change in blood pressure (systolic/diastolic) | Enrollment through Month 18
Amount of change and percent change in blood pressure (systolic/diastolic) | Enrollment through Month 24
Amount of change and percent change in blood pressure (systolic/diastolic) | Enrollment through Month 30
Amount of change and percent change in blood pressure (systolic/diastolic) | Enrollment through Month 36 (or withdrawal from the study)
Occurrence of adverse events | Enrollment through Month 36
Occurrence of cerebral or cardiorenovascular events in the febuxostat group during the study period by febuxostat dose | Enrollment through Month 36
Occurrence of cerebral or cardiorenovascular events in the non-febuxostat group during the study period by use of allopurinol | Enrollment through Month 36

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Ogawa, Study Chair — Department of Cardiovascular Medicine, Graduate School of Medical Sciences, Kumamoto University
Locations (140):
- Japan (140):
  - Hiramitsu Heart Clinic, Nagoya, Aichi-ken
  - Ogawa-naika Clinic, Nagoya, Aichi-ken
  - Shakaiiryohoｊin Koｊunkai Daido Hospital, Nagoya, Aichi-ken
  - Honjo Daiichi Hospital, Yurihonjō, Akita
  - Iriyouhoujin Siyadan Yanagisawakai Yanagisawaiin, Matsudo, Chiba
  - Matsuno Medical Clinic, Iyo-gun, Ehime
  - Ishite Matsumoto Naika Junkanki Clinic, Matsuyama, Ehime
  - Ehime Medical CO-OP Izumigawa Clinic, Niihama, Ehime
  - Hanaoka IC Clinic, Buzen, Fukuoka
  - Otonari Clinic, Chikushino-shi, Fukuoka
  - Saku Hospital, Fukuoka, Fukuoka
  - Tohaya Iin, Fukuoka, Fukuoka
  - Medical Cooperation Toseikai Goto Clinic, Kitakyushu, Fukuoka
  - ONGA NAKAMA Medical Association ONGA Hospital, Onga-gun, Fukuoka
  - Southern Tohoku Research Institute For Neuroscience Southern Tohoku Medical Clinic, Kōriyama, Fukushima
  - Iryohojin Shadan Seijinkai Kawade Iin, Gifu, Gifu
  - Kawai Naika Clinic, Gifu, Gifu
  - Miwa Clinic: Gastroenterology Hepatology, Gifu, Gifu
  - Sagou Clinic, Gifu, Gifu
  - Sasaki Clinic, Gifu, Gifu
  - Takai Clinic, Gifu, Gifu
  - Takeda Clinic, Gifu, Gifu
  - Totani Medical Clinic, Gifu, Gifu
  - Noda Clinic, Ibi, Gifu
  - Sunomata Clinic, Ōgaki, Gifu
  - Tsurugaya Hospital, Isesaki, Gunma
  - Nakano Clinic, Shibukawa, Gunma
  - Iryouhoujinn Makikai Makibyouinn, Takasaki, Gunma
  - Shigenobu Clinic, Miyoshi, Hiroshima
  - Keiyukai Yoshida Hospital, Asahikawa, Hokkaido
  - Matsui Naika Clinic, Asahikawa, Hokkaido
  - Omiya Clinic, Asahikawa, Hokkaido
  - Miyanomori Memorial Hospital, Sapporo, Hokkaido
  - Okamoto Naika Clinic, Sapporo, Hokkaido
  - River Side Clinic, Sapporo, Hokkaido
  - Katsuya Iin, Amagasaki, Hyōgo
  - Kousei Hospital, Himeji, Hyōgo
  - Nakatani Hospital, Himeji, Hyōgo
  - Harima Clinic, Kakogawa, Hyōgo
  - Kusunose Surgery Clinic, Kobe, Hyōgo
  - Yamaki Medical Clinic, Hitachi-Naka, Ibaraki
  - Shika Clinic, Hakui, Ishikawa-ken
  - Yanagi Medical Clinic, Hakusan, Ishikawa-ken
  - Kakuda Iin, Kahoku, Ishikawa-ken
  - Dr Hayakawa's Family Clinic, Kanazawa, Ishikawa-ken
  - Wakasa Medical Clinic, Kanazawa, Ishikawa-ken
  - Okyozuka Clinic, Nonoichi, Ishikawa-ken
  - Matsuoka Clinic, Takamatsu, Kagawa-ken
  - Ori Clinic, Ashigarakami, Kanagawa
  - Iroden Clinic, Kamakura, Kanagawa
  - Nagasu Clinic, Kamakura, Kanagawa
  - Shohei Clinic, Kamakura, Kanagawa
  - Kamegaya Clinic, Kawasaki, Kanagawa
  - Kobayashi Hospital, Odawara, Kanagawa
  - Hakuai Iin, Sagamihara, Kanagawa
  - Yamamoto Clinic, Sagamihara, Kanagawa
  - International Goodwill Hospital, Yokohama, Kanagawa
  - Kikuchi Clinic, Yokohama, Kanagawa
  - Shimokurata Heart Clinic, Yokohama, Kanagawa
  - Tani Clinic Internal Medicine, Allergology & Rheumatology, Yokohama, Kanagawa
  - Tsurumi Chuo Clinic, Yokohama, Kanagawa
  - Yamagami Naika, Yokohama, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokohama Sotetsu bldg Clinic of Internal Medicine, Yokohama, Kanagawa
  - Shimamoto Hospital, Kochi, Kochi
  - Toihata Naika, Aso, Kumamoto
  - Omori Iin, Kōshi, Kumamoto
  - Honjo Internal Medicine Hospital, Kumamoto, Kumamoto
  - Jinnouchi Clinic Diabetes Care Center, Kumamoto, Kumamoto
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Maki Cardiovascular Clinic, Kumamoto, Kumamoto
  - Otsuka Hospital, Kumamoto, Kumamoto
  - Suizenji Touya Hospital, Kumamoto, Kumamoto
  - TERAO Hospital, Kumamoto, Kumamoto
  - Kan Kaimeido Clinic, Tamana, Kumamoto
  - Matsuo Clinic, Tamana, Kumamoto
  - Miyagi clinic cardiovascular medicine, Yatsushiro, Kumamoto
  - Isoda Internal Medical Clinic, Kyoto, Kyoto
  - Koseikai Clinic, Kyoto, Kyoto
  - Takenaka Clinic, Kyoto, Kyoto
  - Iwasaki Hospital, Tsu, Mie-ken
  - Yokota Naika, Miyazaki, Miyazaki
  - Eto Clinic, Nichinan, Miyazaki
  - Kawano Clinic, Nichinan, Miyazaki
  - Miyata Naika Iin, Nobeoka, Miyazaki
  - Nara Medical University Hospital, Kashihara, Nara
  - Ote Clinic of Internal, Sakurai, Nara
  - Uchiyama Clinic, Jōetsu, Niigata
  - Maeda Medical Clinic, Niigata, Niigata
  - Hospital, University of the Ryukyus, Nakagami, Okinawa
  - Nishimura Clinic, Fujiidera, Osaka
  - Ikeda Clinic, Higashiosaka, Osaka
  - Kanazawa Clinic, Izumi, Osaka
  - Akioka Clinic, Osaka, Osaka
  - Kinugawa Cardiology Clinic, Osaka, Osaka
  - Kondo Clinic, Osaka, Osaka
  - Kubota Clinic, Osaka, Osaka
  - Matsushita Medical Clinic, Osaka, Osaka
  - Nanko Clinic, Osaka, Osaka
  - Seo Heart Clinic, Osaka, Osaka
  - Watanabe Iin, Osaka, Osaka
  - Hayashi Medical Clinic, Sakai, Osaka
  - Matsuo Clinic, Yao, Osaka
  - Enomoto Clinic, Ageo, Saitama
  - Saitama Medical Center, Kawagoe, Saitama
  - Iryohojin Hogi sinryojyo, Kawaguchi, Saitama
  - Okuaki Clinic, Kawaguchi, Saitama
  - Tokutake Iin, Kawaguchi, Saitama
  - Medical Corporation Shibuya Clinic, Kumagaya, Saitama
  - Harada Medical Clinic, Shizuoka, Shizuoka
  - Shizuoka Municipal Hospital, Shizuoka, Shizuoka
  - Waki Riichiro Clinic, Shizuoka, Shizuoka
  - Ota Clinic, Awa, Tokushima
  - Minami National Health Insurance Hospital Of Minami Town, Kaifu-gun, Tokushima
  - Sekishinkan Hospital, Komatsushimachō, Tokushima
  - Tanaka Clinic, Myozai-gun, Tokushima
  - Itsumo Smile Clinic, Tokushima, Tokushima
  - Harada Clinic, Adachi-ku, Tokyo
  - Johoku Clinic, Adachi-ku, Tokyo
  - Moritani Clinic, Bunkyo-ku, Tokyo
  - Nishimura Memorial Hospital, Edogawa-ku, Tokyo
  - Hosoda-Clinic, Katsushika-ku, Tokyo
  - Okuda clinic, Kita-ku, Tokyo
  - Tenjinmae Clinic, Mitaka, Tokyo
  - Daiba Shinryojo, Nakano-ku, Tokyo
  - Kurumatani Clinic, Nerima-ku, Tokyo
  - Oono Iin, Nerima-ku, Tokyo
  - Sugawara Clinic, Nerima-ku, Tokyo
  - Baba Iin, Nishitōkyō, Tokyo
  - Miyahara Clinic, Ōta-ku, Tokyo
  - Taguchi Clinic, Shinagawa-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo
  - Kobayashi Clinic, Suginami-ku, Tokyo
  - Tominaga Clinic, Tachikawa, Tokyo
  - Kirino Clinic, Toshima-ku, Tokyo
  - Yamada Clinic, Toshima-ku, Tokyo
  - Shimasaki Clinic, Yamagata, Yamagata
  - Ayame Medical Clinic, Shimonoseki, Yamaguchi
  - Matuda Clinic, Shimonoseki, Yamaguchi
  - Kuroda Iin, Ōtsuki, Yamanashi Pref.

REFERENCES:
- [Derived] Sugawara M, Kojima S, Hisatome I, Matsui K, Uchiyama K, Yokota N, Tokutake E, Wakasa Y, Hiramitsu S, Waki M, Jinnouchi H, Kakuda H, Hayashi T, Kawai N, Mori H, Tsujita K, Ohya Y, Kimura K, Saito Y, Ogawa H; Febuxostat for Cerebral and CaRdiorenovascular Events PrEvEntion StuDy (FREED) investigators. Impacts of Febuxostat on Cerebral and Cardiovascular Events in Elderly Patients with Hyperuricemia: Post Hoc Analysis of a Randomized Controlled Trial. Clin Pharmacol Ther. 2024 Jun;115(6):1358-1364. doi: 10.1002/cpt.3217. Epub 2024 Feb 23. PMID 38389505
- [Derived] Kojima S, Uchiyama K, Yokota N, Tokutake E, Wakasa Y, Hiramitsu S, Waki M, Jinnouchi H, Kakuda H, Hayashi T, Kawai N, Sugawara M, Mori H, Tsujita K, Matsui K, Hisatome I, Ohya Y, Kimura K, Saito Y, Ogawa H; Febuxostat for Cerebral and CaRdiorenovascular Events PrEvEntion StuDy (FREED) investigators. C-reactive Protein Levels and Cardiovascular Outcomes After Febuxostat Treatment in Patients with Asymptomatic Hyperuricemia: Post-hoc Analysis of a Randomized Controlled Study. Cardiovasc Drugs Ther. 2023 Oct;37(5):965-974. doi: 10.1007/s10557-022-07347-7. Epub 2022 Jun 1. PMID 35648242
- [Derived] Kojima S, Uchiyama K, Yokota N, Tokutake E, Wakasa Y, Hiramitsu S, Waki M, Jinnouchi H, Kakuda H, Hayashi T, Kawai N, Sugawara M, Mori H, Tsujita K, Matsui K, Hisatome I, Ohya Y, Kimura K, Saito Y, Ogawa H; Febuxostat for Cerebral and Cardiorenovascular Events Prevention Study (FREED) investigators. Optimal uric acid levels by febuxostat treatment and cerebral, cardiorenovascular risks: post hoc analysis of a randomized controlled trial. Rheumatology (Oxford). 2022 May 30;61(6):2346-2359. doi: 10.1093/rheumatology/keab739. PMID 34605897
- [Derived] Kojima S, Matsui K, Hiramitsu S, Hisatome I, Waki M, Uchiyama K, Yokota N, Tokutake E, Wakasa Y, Jinnouchi H, Kakuda H, Hayashi T, Kawai N, Mori H, Sugawara M, Ohya Y, Kimura K, Saito Y, Ogawa H. Febuxostat for Cerebral and CaRdiorenovascular Events PrEvEntion StuDy. Eur Heart J. 2019 Jun 7;40(22):1778-1786. doi: 10.1093/eurheartj/ehz119. PMID 30844048
- [Derived] Kojima S, Matsui K, Ogawa H, Jinnouchi H, Hiramitsu S, Hayashi T, Yokota N, Kawai N, Tokutake E, Uchiyama K, Sugawara M, Kakuda H, Wakasa Y, Mori H, Hisatome I, Waki M, Ohya Y, Kimura K, Saito Y; Febuxostat for Cerebral and Cardiorenovascular Events Prevention Study (FREED) investigators. Rationale, design, and baseline characteristics of a study to evaluate the effect of febuxostat in preventing cerebral, cardiovascular, and renal events in patients with hyperuricemia. J Cardiol. 2017 Jan;69(1):169-175. doi: 10.1016/j.jjcc.2016.02.015. Epub 2016 Apr 20. PMID 27005768